CLINICAL TRIAL: NCT04980742
Title: Perioperative Risk Factors of Outcomes for Cardiac Surgery: A Retrospective Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: 2017-111
Record Dates: First submitted 2020-08-23; First posted 2021-07-28 (Actual); Last update posted 2021-07-28 (Actual); Status verified 2020-08

CONDITIONS: Post-cardiac Surgery; Blood Transfusion Complication; Prognosis
MeSH Terms: conditions — Transfusion Reaction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: acute normovolemic hemodilution — acute normovolemic hemodilution

SUMMARY:
Based on a review of about 10,000 patients undergoing cardiac surgery under CPB in West China Hospital of Sichuan University and the Second Affiliated Hospital of Zhejiang University, we try to evalute the effect of blood transfusion on outcomes in cardiac surgery.

DETAILED DESCRIPTION:
Based on a review of about 10,000 patients undergoing cardiac surgery under CPB in West China Hospital of Sichuan University and the Second Affiliated Hospital of Zhejiang University, the following results were obtained:

1. Perioperative risk factors of death and complications of different organ systems after cardiac surgery, providing evidence for early prevention and intervention;
2. Risk factors of blood transfusion risk were analyzed to provide ideas for reducing intraoperative blood transfusion;
3. The relationship between hemoglobin and complications after heart surgery was explored to provide a factual basis for the development of blood transfusion indications for such patients

ELIGIBILITY:
Inclusion Criteria:

* The patients in the west China hospital of sichuan university (July 01, 2011, solstice during June 30, 2017) and the second affiliated hospital of zhejiang university (September 01, 2013, solstice, June 30, 2017) have cardiac surgery under Cardiopulmonary bypass (CPB)

Exclusion Criteria:

* No

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients in the west China hospital of sichuan university (July 01, 2011, solstice during June 30, 2017) and the second affiliated hospital of zhejiang university (September 01, 2013, solstice, June 30, 2017) have cardiac surgery under Cardiopulmonary bypass (CPB)
Sampling Method: Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2017-07-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
mortality | 28 days after surgery
  all-cause death

CONTACTS AND LOCATIONS:
Overall Officials: Min Yan, doctor, Study Chair — The Second Affiliated Hospital of Zhejiang University Medical College
Locations (1):
- ANH, Hangzhou, China

IPD SHARING:
Plan to Share IPD: Undecided